CLINICAL TRIAL: NCT02751905
Title: A Phase 1, Open-Label Study to Evaluate the Absorption, Metabolism, and Excretion of [14C]-BIIB074 in Healthy Male Subjects
Brief Title: Absorption, Metabolism, and Excretion Study of BIIB074
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 802HV105
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — vixotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIIB074 (Experimental): Single oral dose on Day 1
  Interventions: Drug: BIIB074

INTERVENTIONS:
Drug: BIIB074 — Administered orally as specified in treatment arm
  Other Names: CNV1014802

SUMMARY:
The primary objectives of the study are: To determine the mass balance and routes of elimination of BIIB074 and its known metabolites following administration of a single oral dose of BIIB074 in healthy male participants and To describe the pharmacokinetics (PK) of BIIB074 and its known metabolites and the disposition profiles of total radioactivity in whole blood and plasma following a single oral dose. The secondary objectives of this study are: To assess the safety and tolerability of BIIB074 in healthy participants and To identify and characterize any additional metabolites of BIIB074 in plasma, urine, and feces.

ELIGIBILITY:
Key Inclusion Criteria:

* All subjects must practice effective contraception during the study and be willing and able to continue contraception for 90 days after the administration of study treatment.
* Must be in good health as determined by the Investigator, based on medical history and screening evaluations.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* Previous exposure to BIIB074.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen, make the subject unsuitable for enrollment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Urinary amount excreted per sampling interval (Aeu) | 12 hours prior to dosing up to Day 9
Fecal amount excreted per sampling interval (Aef) | Prior to dosing up to Day 9
Cumulative urinary amount excreted per sampling interval (Cum Aeu) | 12 hours prior to dosing up to Day 9
Cumulative fecal amount excreted per sampling interval (Cum Aef) | Prior to dosing up to Day 9
Percentage of radioactive urinary dose excreted per sampling interval (%Feu) | 12 hours prior to dosing up to Day 9
Percentage of radioactive fecal dose excreted per sampling interval (%Fef) | Prior to dosing up to Day 9
Cumulative percentage of radioactive urinary dose excreted per sampling interval (Cum %Feu) | 12 hours prior to dosing up to Day 9
Cumulative percentage of radioactive fecal dose excreted per sampling interval (Cum %Fef) | Prior to dosing up to Day 9
Urinary amount of BIIB074 and its known metabolites excreted per sampling interval (Aeu) | 12 hours prior to dosing up to Day 9
Cumulative urinary amount of BIIB074 and its known metabolites excreted per sampling interval (Cum Aeu) | 12 hours prior to dosing up to Day 9
Percentage of BIIB074 dose excreted per sampling interval (%Feu) | 12 hours prior to dosing up to Day 9
Cumulative percentage of BIIB074 dose excreted (Cum %Feu) | 12 hours prior to dosing up to Day 9
Maximum observed concentration (Cmax) | 2 hours post dose up to Day 9
Time to reach Cmax (Tmax) | 2 hours post dose up to Day 9
Area under the concentration-time curve from time 0 to time of the last measurable drug concentration (AUC0-t) | 2 hours post dose up to Day 9
Area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf) | 2 hours post dose up to Day 9
Terminal elimination half-life (t1/2) | 2 hours post dose up to Day 9
Apparent total body clearance (CL/F) | 2 hours post dose up to Day 9
Apparent volume of distribution (Vd/F) | 2 hours post dose up to Day 9
Renal clearance (CLR) | 2 hours post dose up to Day 9
Metabolite-to-parent ratio at Cmax (MRCmax) | 2 hours post dose up to Day 9
Metabolite-to-parent ratio in AUC (MRAUC) | 2 hours post dose up to Day 9

SECONDARY OUTCOMES:
Number of participants experiencing adverse events (AEs) and serious adverse events (SAEs) | Up to Day 9
Number of participants with clinically significant vital sign abnormalities | Up to Day 9
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | Up to Day 9
Number of participants with clinically significant laboratory assessment abnormalities | Up to Day 9
Radioactivity profiles in plasma, urine and feces | Up to Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Madison, Wisconsin, United States